CLINICAL TRIAL: NCT04862507
Title: Improving Low Alberta Stroke Program Early ct Score Stroke Thrombectomy
Brief Title: Improving Low ASPECTS Stroke Thrombectomy
Acronym: I-LAST
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University of Kaiserslautern (Other); University Hospital Muenster (Other); University of Rostock (Other); University Hospital, Basel, Switzerland (Other); Charite University, Berlin, Germany (Other); Klinikum Bremen-Mitte, gGmbH (Other)
Responsible Party: Principal Investigator, Gabriel Broocks, Assistant Professor, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: I-LAST
Record Dates: First submitted 2021-04-13; First posted 2021-04-28 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Patients with an ASPECTS of 0-5 on baseline neuroimaging undergoing thrombectomy: acute stroke patients treated with endovascular treatment combined with thrombolysis or without previous thrombolysis Intervention.
  Interventions: Other: Telephone call on day 90; Diagnostic Test: Quantification of lesion water uptake by CT densitometry
- Stroke Patients with an ASPECTS of 0-5 on baseline neuroimaging not undergoing thrombectomy: acute stroke patients treated with or without thrombolysis
  Interventions: Other: Telephone call on day 90; Diagnostic Test: Quantification of lesion water uptake by CT densitometry

INTERVENTIONS:
Other: Telephone call on day 90 — telephone call on day 90 to assess the primary outcome (mRs 90)
Diagnostic Test: Quantification of lesion water uptake by CT densitometry — Retrospective quantification of lesion water uptake by CT densitometry in admission and follow-up imaging

SUMMARY:
Improving Low ASPECTS Stroke Thromectomy (I-LAST) is an academic, independent, prospective, multicenter, observational registry study. Consecutive patients treated with endovascular stroke treatment will be enrolled in German stroke centers. Patients receive regular care and data will be collected as part of clinical routine. Baseline clinical and procedural information as well clinical follow-up information during in-hospital stay, and up to 90 days of stroke onset are collected. Data collected include demographics, National Institute of Health Stroke Scale (NIHSS) on admission, pre-treatment ASPECTS, information on timing and success of interventional treatment, procedural complications, intracranial hemorrhage, and functional outcome. Advanced imaging biomarkers will be tested and validated aiming to improve treatment selection and outcome prediction of patients presenting with extensive baseline infarction.

DETAILED DESCRIPTION:
This study aims to investigate the role of advanced imaging biomarkers in patients with large early infarct, in particular quantitative lesion water uptake (Minnerup et al. Annals of Neurology 2016), arterial and venous collateral circulation (Faizy et al. Radiology 2021), and multivariate CTP-derived parameters (Kemmling et al. JCBFM 2015). The goal is to use these imaging biomarkers as specific selection criterion to predict clinical benefit after reperfusion despite extensive baseline infarct lesions, also as a method of monitoring adjuvant neuroprotective agents after reperfusion therapy (for instance anti-edematous medication).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* ASPECTS of 0-5
* Confirmed diagnosis of persistent occlusion of terminal carotid artery, middle cerebral artery (M1 or M2), or basilar artery consistent with symptoms
* Age >18 years
* Ethic approval in process

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute stroke patients with the clinical diagnosis of acute ischemic stroke with a ASPECTS 0f 0-5 on baseline imaging; Age >18 years
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
modified ranking scale on day (mRs) day 90 | 90 days
  mRs: modified ranking scale; the scale is a commonly used measurement for the degree of disability or dependence in the daily activities of people who have suffered a stroke; scale range 0-6, with 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead. publication: van Swieten J, Koudstaal P, Visser M, Schouten H, et al. (1988). "Interobserver agreement for the assessment of handicap in stroke patients". Stroke. 19 (5): 604-607. doi:10.1161/01.str.19.5.604.

SECONDARY OUTCOMES:
Ischemic lesion water uptake on admission | 0-24 hours after symptom onset
  Ischemic lesion water uptake is a CT based quantitative imaging biomarker to assess ischemic edema based on densitometry
Ischemic lesion water uptake on follow-up imaging | 24-48 hours after admission
  Ischemic lesion water uptake is a CT based quantitative imaging biomarker to assess ischemic edema based on densitometry

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (7):
  - Charite University Berlin, Berlin
  - Hospital Bremen-Mitte, Bremen
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Westpfalzklinikum, Kaiserslautern
  - University Hospital Marburg, Marburg
  - University Münster, Münster
  - University Rostock, Rostock
- University Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request.

REFERENCES:
- [Derived] Broocks G, Meyer L, Elsayed S, McDonough R, Bechstein M, Faizy TD, Sporns P, Schon G, Minnerup J, Kniep HC, Hanning U, Barow E, Schramm P, Langner S, Nawabi J, Papanagiotou P, Wintermark M, Lansberg MG, Albers GW, Heit JJ, Fiehler J, Kemmling A; I-LAST Investigators. Association Between Net Water Uptake and Functional Outcome in Patients With Low ASPECTS Brain Lesions: Results From the I-LAST Study. Neurology. 2023 Feb 28;100(9):e954-e963. doi: 10.1212/WNL.0000000000201601. Epub 2022 Nov 22. PMID 36414425